CLINICAL TRIAL: NCT02126644
Title: Phase 2 Study of the Efficacy and Safety of a Single 70% Glycolic Acid Peel With Vitamin C for the Treatment of Photoaging
Brief Title: The Efficacy and Safety of a Single 70% Glycolic Acid Peel With Vitamin C for the Treatment of Photoaging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/01229
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Photoaging
Keywords: Photoaging; 70% glycolic acid peel
MeSH Terms: interventions — glycolic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Single arm of 10 patients - efficacy and safety assessed pre and post peel
  Interventions: Drug: 70% glycolic acid

INTERVENTIONS:
Drug: 70% glycolic acid

SUMMARY:
Our study involves the evaluation of a high potency peel in its efficacy for skin rejuvenation in the treatment of photoaging. This chemical peel regime is a high potency peel 70% glycolic acid combined with vitamin C that is purported to provide a good balance between yielding results and patient safety.

AIM We aim to qualitatively evaluate its efficacy and safety profile.

Our hypothesis is that a single peel of 70% glycolic acid combined with vitamin C will result in improvement of the features of photoaging with few side effects.

DETAILED DESCRIPTION:
1. Assessment of photoaging to compare using photography A and E - for static analysis.

   For each element from ii to xi, a rating of nil (0), mild (l), moderate (2), and severe (3) for each category was made by the same evaluating physician.

   i. Physician VAS scale - assessment of wrinkles prepeel, post peel (Score 1 -10).

   ii.Fine peri-orbital wrinkles (less than 1 mm in width or depth) (FPW); iii.Course peri-orbital wrinkles (greater than 1 mm in width and depth) (CPW); iv.Upper lip wrinkles (ULW); v.Lower lip wrinkles (LLW); vi.Melasma defined as blotchy, brown, epidermal macules with indistinct margins; vii.Solar lentigines defined as dark brown macules with distinct margins measuring from 3 to 10 mm; viii.Solar keratoses defined as diffuse erythema with keratotic adherent scaling; ix.Guttate hypomelanosis defined as localized macules of absent melanin measuring from 3 to 10 mm in diameter; x.Poikiloderma defined as a symmetrical reddish-brown pigmentation of the neck, typically sparing the sub-mental area;

   The totaling of the scores of the above parameters will form a prepeel score. This will be compared against the patient's score post peel - we expect to find an improvement.
2. Safety profile assessment

   * redness, swelling, oozing, hyperpigmentation, scarring
   * each of the 5 parameters will be scored from 0 -3, none, mild, moderate, severe
   * this will serve as a safety assessment.

ELIGIBILITY:
Inclusion Criteria:

Photoaging Grade 2-4 (face) Skin type I - IV

Exclusion Criteria:

* Pregnancy, breast feeding Active dermatitis on the face, rosacea, allergic rhinitis, herpes Known hypersensitivity Previous Keloids Laser ablative procedures within the last one month Chemical Peels in the last 6 months Used oral retinoids in the last 6 months Used topical retinoids in the past one week Used Scrub, Alpha Hydroxy Acid, skin irritant for the past 24h Presence of facial warts, fungal infections Photoallergies Prior poor reaction to a chemical peel Radiotherapy Skin type V and VI

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of Parameters for Photoaging | 3 months
  i. Physician VAS scale - Score 1 -10. ii.Fine peri-orbital wrinkles iii.Course peri-orbital wrinkles; iv.Upper lip wrinkles (ULW); v.Lower lip wrinkles (LLW); vi.Melasma vii.Solar lentigines viii.Solar keratoses ix.Guttate hypomelanosis x.Poikiloderma
  The totaling of the scores of the above parameters will form a prepeel score. This will be compared against the patient's score post peel - we expect to find an improvement.
Safety Assessment | 3 months
  Safety profile assessment
  * redness, swelling, oozing, hyperpigmentation, scarring
  * each of the 5 parameters will be scored from 0 -3, none, mild, moderate, severe

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore